CLINICAL TRIAL: NCT01408628
Title: The I-KAN Study: Internet Initiation of Insulin for Type 2 Diabetes in Kansas
Brief Title: The I-KAN Study: Internet Insulin Education for Kansans
Acronym: I-KAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Robbins, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David Robbins, MD, Professor and Director KU Diabetes Institute, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 12634; 1R34DK089444-01A1 (NIH)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2015-05-18 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Internet Insulin Education (Experimental): Single arm study; intervention represented by subjects' participation in 4 synchronous ("live") interactive Internet classes.
  Interventions: Behavioral: Internet Insulin Education

INTERVENTIONS:
Behavioral: Internet Insulin Education — Offer and assess the safety and effectiveness of a synchronous ("live") interactive 4-week Internet course designed to teach groups of type 2 diabetic patients to safely administer basal insulin without significant support from their usual source of diabetic management and to self-adjust the dose to achieve an HbA1c of < 7.0% using an established treat-to-target algorithm.

SUMMARY:
The primary purpose of the study is demonstration that teaching insulin management in small groups of type 2 diabetes patients in 4 weekly "live" Internet sessions is safe and provides an important resource for rural diabetes care providers who may otherwise, because of lack of time or staff, not be able to put patients on insulin who need it.

DETAILED DESCRIPTION:
The proposed project will test in a limited number of rural and semi-rural sites in the state of Kansas an innovative model of synchronous ("live") Internet initiation and intensification of once daily basal insulin glargine or detemir in type 2 diabetic patients that can be deployed statewide in a subsequent larger study (R18). The study's specific aims are to 1) develop a synchronous ("live") interactive Internet-administered course designed to teach groups of type 2 diabetic patients to safely administer basal insulin without significant support from their usual source of diabetic management and to self-adjust the dose to achieve a HbA1c < 7.0% using a treat-to-target algorithm; and 2) to assess for the Internet patients selected clinical and psychometric outcomes. These will include HbA1c, frequency and severity of hypoglycemia, psychological resistance to insulin treatment, diabetes quality of life, and treatment satisfaction. The study builds upon the findings of the Treat-to-Target and INITIATE trials, as well as on successful Internet interventions for weight management, and both lays the conceptual foundation and gathers the expertise to successfully apply for the R18, which will have as primary aims addressing of delays to insulin therapy documented in the DAWN study and cost effectiveness analysis of the Internet intervention. The study hopes to show that Internet teaching of basal insulin therapy is comparable to traditional insulin management with respect to safety and effectiveness as measured against expected (published) results for frequency of hypoglycemia and percent of patients reaching target. Psychometric outcomes are exploratory - and hypothesis generating with respect to the subsequent R18 application.

ELIGIBILITY:
Inclusion Criteria:

* T2DM, meets provider criteria for insulin initiation; starting or having started insulin treatment no longer than six months prior to enrollment OR has not yet committed to starting insulin but has agreed to participate in the education
* broadband Internet and experience with logging into a password-protected site (e.g., eCommerce or social networking);
* ability to purchase or otherwise acquire glargine/detemir insulin and testing supplies.

Exclusion Criteria:

* Use of oral glucocorticoids or second generation anti-psychotics;
* previous use of self-administered insulin more than six months prior to enrollment;
* gestational diabetes or other endocrine conditions causing hyperglycemia; treatment for a malignant condition other than basal cell carcinoma in situ within prior two years;
* renal insufficiency (AST/ALT >2 or concurrent liver disease except NASH);
* pregnant or planning to become pregnant within 6 months;
* HbA1c < 7.0% or ongoing weight loss or persistent fasting hyperglycemia > 250 mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Robbins, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Consented
Arm/Group | Internet Insulin Education
Started | 51
Completed | 39
Not Completed | 12
Not completed — Withdrawal by Subject | 12
Period: Started Classes/Intervention
Arm/Group | Internet Insulin Education
Started | 39
Completed | 39
Not Completed | 0
Period: Completed 6 Month Follow-Up
Arm/Group | Internet Insulin Education
Started | 39
Completed | 25
Not Completed | 14
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Internet Insulin Education
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.67 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 51
A1c Baseline [Mean (Standard Deviation); unit: Percentage (glycosolated hemoglobin)] | 8.61 (1.63)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Hypoglycemia
Description: Hypoglycemia was defined in the study as either a blood glucose reading <70 mg/dL or symptomatic to the patient/subject.
Time Frame: 6-month follow up period following the Internet Intervention
Population: Subjects who both completed the Internet intervention AND the 6 months of follow up
Measure: Mean (Standard Deviation); unit: incidents per person-year
Groups:
- Internet Insulin Education: Internet Insulin Education: Offer and assess the safety and effectiveness of a synchronous ("live") interactive 4-week Internet course designed to teach groups of type 2 diabetic patients to safely administer basal insulin without significant support from their usual source of diabetic management and to self-adjust the dose to achieve an HbA1c of ≤ 7.0% using an established treat-to-target algorithm.
Arm/Group | Internet Insulin Education
Number analyzed (Participants) | 25
incidents per person-year | 6.88 (11.20)

2. Secondary Outcome: Change in HbA1c
Description: Change in HbA1c (average measure of the % of glycosolated hemoglobin in the blood over the past 3 months) from baseline to end of follow up period.
Time Frame: Change from Baseline through Month 6 of follow-up period
Population: Subjects who both completed the Internet intervention and the six months of follow up
Measure: Mean (Standard Deviation); unit: percentage of glycosolated hemoglobin
Arm/Group | Internet Insulin Education
Number analyzed (Participants) | 25
percentage of glycosolated hemoglobin | -1.33 (1.44)

3. Secondary Outcome: Severity of Self-reported Hypoglycemia
Description: Severity was defined by the scale used by the DCCT: grade 1 - subject was able to recognize and treat appropriately without assistance; grade 2 - subject required help from another person either to recognize or recognize/treat; grade 3 - subject required injection of glucagon or treatment in ER
Time Frame: 6 Months
Population: Subjects who completed both the Internet intervention and the 6 months of follow up
Measure: Number; unit: incidents (count)
Arm/Group | Internet Insulin Education
Number analyzed (Participants) | 25
incidents (count)
  Grade 1 | 141
  Grade 2 | 1
  Grade 3 | 0

ADVERSE EVENTS:
Time Frame: 6 month follow up period post Internet intervention
Description: Adverse events were defined as hypoglycemic events (either a blood glucose reading <70 or symptomatic hypoglycemia). Our formal data collection included only hypoglycemia as an adverse event. Subjects continued to see their primary care providers throughout the study for any medical issues unrelated to the intervention.
Arm/Group | Internet Insulin Education
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 10/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Internet Insulin Education (N=39)
Hypoglycemia (Endocrine disorders) | 10 (142) — Of the 51 people enrolled on the study, 39 continued on to the intervention phase. The 12 people that withdrew before the intervention phase were not at risk for hypoglycemia since they had not started insulin.

LIMITATIONS AND CAVEATS:
This was a pilot study designed to compare rates of hypoglycemia among Internet managed type 2 patients to those from large clinical trials. It was not a placebo controlled trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes